CLINICAL TRIAL: NCT05419973
Title: Vitamin D Levels in Umbilical Cord and It's Impact on Infant and Children's Health (VITADi Study)
Acronym: VITADi
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, dr. Sri Hardiyanti Putri, Sp.A, Principal Investigator, Pediatrician, Teaching Staff at Pediatric Department Hasanuddin University, Hasanuddin University
Other Study IDs: UH22030108
Record Dates: First submitted 2022-06-11; First posted 2022-06-15 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D in Infants
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Women: Women in third semester of pregnancy who are willing to include their babies as samples for the next study, no history of abortion, and not suffering from hypertension and preeclampsia.
  Interventions: Other: Anthropometric measurement for pregnant women; Other: Blood sampling
- Infants: Babies born from mothers who are willing to be included in the study, aterm, with birth weight more than 2500 grams. No congenital abnormalities at birth and no acute infection at birth.
  Interventions: Other: Anthropometric measurement for infants; Other: Blood sampling

INTERVENTIONS:
Other: Anthropometric measurement for pregnant women — Weight, length, upper arm circumference
  Groups: Pregnant Women
Other: Anthropometric measurement for infants — birth weight, length, head circumference, nutritional status
  Groups: Infants
Other: Blood sampling — 3 ml of blood will be taken, 1,5 ml each to measure the complete blood count, and other 1,5 ml to measure ferritin, Fe serum, vitamin D levels, vitamin D receptors, IL-6 and IL-10.

SUMMARY:
This study is a cohort study that aims to assess the relationship between Vitamin D Levels in infant and the risk of anemia, atopic dermatitis, diarrhea and cardiovascular disorders in newborn. The subjects of this study are 100 women who met the inclusion criteria, which are in their third trimester of pregnancy and agree to be included in this study. These subjects then will be examined for their weight using standardized CEBA digital scale, height, upper arm circumference, and blood sampling will also be done to these women to measure their vitamin D levels, calcium, parathyroid hormone, ferritin, Fe serum, IL-16, IL-10. When subjects give birth, the babies will also be included in this study. Anthropometric examination will also be done on the babies, to measure their birth weight, birth length, and head circumference. Blood samples will also be taken from their umbilical cord to assess their complete blood count, ferritin, Fe serum, vitamin D levels, vitamin D receptors, IL-6 and IL-10. All subjects then will be monitored, and home visits will be done when the babies reach 3 months old and 6 months old. An assessment of the incidence of diarrhea, atopic dermatitis, and an assessment of cardiovascular disorders (checking pulse and blood pressure) will be carried out during the visit. At the end of the study, venous blood sampling will be taken to see levels of vitamin D, calcium, parathyroid hormone, routine complete blood count, serum Fe, and ferritin, then data analysis is performed.

DETAILED DESCRIPTION:
Participants of this study are women in the third semester of pregnancy, who consented to be included with their babies in this study. Firstly, the parents will be given explanation regarding the study, and informed consent will be signed if they agree to participate. All the pregnant women who met the criteria will be recorded for their name, age, parity, birth and medical history. Anthropometric examination will be done on the pregnant women, to measure weight using standardized CEBA digital scale, height and upper arm circumference. Blood sampling will also be done to measure complete blood count, ferritin, Fe serum, vitamin D levels, calcium, parathyroid hormone, IL-6 and IL-10.

After the subjects give birth, the babies who met the criteria (aterm, birth weight > 2500 grams, with no congenital abnormalities and acute infection at birth) will also be included in this study. Measurement of birth weight, birth length, and head circumference will be carried out along with blood sampling by taking 3 ml of blood from umbilical cord, 1,5 ml each to measure the complete blood count, and other 1,5 ml to measure ferritin, Fe serum, vitamin D levels, vitamin D receptors, IL-6 and IL-10. Subjects will be monitored for 6 months, and two home visits will be done throughout the study at the age of 3 months and 6 months. During the visits, subjects will be measured for their weight, length, head circumference, as well as their nutritional status. Parents and guardians will also be asked questions regarding the incidence of diarrhea, allergic manifestations such as rash, and assessment will be made based on Hanifin Rajka criteria. At the age of 6 months old, blood sampling will be done again by taking 3 ml of the blood, 1,5 ml each to measure the complete blood count, and other 1,5 ml to measure ferritin, Fe serum, vitamin D levels, vitamin D receptors, IL-6 and IL-10.

The collected data then will be grouped based on the purpose and type of data, then univariate analysis and bivariate analysis will be performed. Univariate analysis will describe the characteristics of the basic data, in the form of frequency, mean value, standard deviation, and range. Meanwhile bivariate analysis such as Wilcoxon test will be performed to to analyse data with independent variables with an ordinal/numeric scale, the data are not normally distributed and have different variances. Mann-Whitney test will also be performed test to compare ordinal or numeric scale variables whose data are not normally distributed and have different variances between two unpaired groups.

ELIGIBILITY:
Inclusion Criteria:

* Women in third trimester of pregnancy
* Agree to include their babies in this study

Exclusion Criteria:

* History of abortion
* Suffering from hypertension or preeclampsia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women in third trimester of pregnancy in Makassar, Surabaya, Mataram who are selected during the screening test.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Vitamin D Levels | August 2022 - February 2023
  Measured by blood sample collection

SECONDARY OUTCOMES:
Hemoglobin levels | August 2022 - February 2023
  Measured by blood sample collection
IgE | August 2022 - February 2023
  Measured by blood sample collection
Atopic Dermatitis | August 2022 - February 2023
  Skin rash, itchiness, patchy skin
Diarrhea | August 2022 - February 2023
  Incidence of diarrhea
Hypertension | August 2022 - February 2023
  Blood pressure obtained during visits

CONTACTS AND LOCATIONS:
Overall Officials: Sri Hardiyanti Putri, MD, Principal Investigator — Hasanuddin University
Locations (1):
- Hasanuddin University, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
We are going to share individual participant data that underlie results in this publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: The data will be shared by email sent by the primary investigator

REFERENCES:
- See also: Atkinson, MA, Melamed, ML, Kumar, J., Roy, CN, Miller, ER, 3rd, Furth, SL, & Fadrowski, JJ (2014). Vitamin D, race, and risk for anemia in children. The Journal of pediatrics, 164(1), 153-158.e1. — https://doi.org/10.1016/j.jpeds.2013.08.060
- See also: Cadario, F., Savastio, S., Pozzi, E., Capelli, A., Dondi, E., Gatto, M., Zaffaroni, M., & Bona, G. (2013). Vitamin D status in cord blood and newborns: Ethnic differences. Italian Journal of Pediatrics, 39(1). — https://doi.org/10.1186/1824-7288-39-35
- See also: Cyprian, F., Lefkou, E., Varoudi, K., & Girardi, G. (2019). Immunomodulatory Effects of Vitamin D in Pregnancy and Beyond. Frontiers in Immunology, 10. — https://doi.org/10.3389/fimmu.2019.02739

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT05419973/Prot_SAP_000.pdf